CLINICAL TRIAL: NCT00091793
Title: A Randomized, Double-Blind Study to Evaluate AMG 162 in the Prevention of Postmenopausal Osteoporosis
Brief Title: Study to Evaluate AMG 162 in the Prevention of Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20040132
Record Dates: First submitted 2004-09-17; First posted 2004-09-21 (Estimated); Results first posted 2010-01-26 (Estimated); Last update posted 2010-12-31 (Estimated); Status verified 2010-12

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Osteoporosis; Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- AMG 162 (Experimental): 60 mg/mL denosumab given day 1, month 6, month 12 and month 18
  Interventions: Drug: AMG 162
- Placebo (Placebo Comparator): Placebo given day 1, month 6, month 12 and month 18
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 162 — 60 mg/mL denosumab given day 1, month 6, month 12 and month 18
  Arms: AMG 162
Drug: Placebo — Placebo given at day 1, month 6, month 12 and month 18
  Arms: Placebo

SUMMARY:
This study will determine whether treatment with AMG 162 can prevent lumbar spine bone loss in both early and late postmenopausal women with osteopenia, and to further test the safety and tolerability of AMG 162 in this population.

ELIGIBILITY:
Eligibility Criteria

- Postmenopausal women with Osteopenia (lumbar spine bone mineral density T-score between 1.0 and -2.5)

Max Age: 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2004-08; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Bone HG, Bolognese MA, Yuen CK, Kendler DL, Wang H, Liu Y, San Martin J. Effects of denosumab on bone mineral density and bone turnover in postmenopausal women. J Clin Endocrinol Metab. 2008 Jun;93(6):2149-57. doi: 10.1210/jc.2007-2814. Epub 2008 Apr 1. PMID 18381571
- [Result] Engelke K, Libanati C, Liu Y, Wang H, Austin M, Fuerst T, Stampa B, Timm W, Genant HK. Quantitative computed tomography (QCT) of the forearm using general purpose spiral whole-body CT scanners: accuracy, precision and comparison with dual-energy X-ray absorptiometry (DXA). Bone. 2009 Jul;45(1):110-8. doi: 10.1016/j.bone.2009.03.669. Epub 2009 Apr 2. PMID 19345291
- [Derived] Bone HG, Bolognese MA, Yuen CK, Kendler DL, Miller PD, Yang YC, Grazette L, San Martin J, Gallagher JC. Effects of denosumab treatment and discontinuation on bone mineral density and bone turnover markers in postmenopausal women with low bone mass. J Clin Endocrinol Metab. 2011 Apr;96(4):972-80. doi: 10.1210/jc.2010-1502. Epub 2011 Feb 2. PMID 21289258
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Denosumab 60 mg Q6M | Placebo
Started | 166 | 166
Completed | 142 | 144
Not Completed | 24 | 22
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 10 | 15
Not completed — Ineligibility determined | 2 | 0
Not completed — Lost to Follow-up | 7 | 5
Not completed — Noncompliance | 2 | 0
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab 60 mg Q6M | Placebo | Total
Number analyzed (Participants) | 166 | 166 | 332
Age Continuous [Mean (Standard Deviation); unit: Years] | 59.8 (7.4) | 58.9 (7.5) | 59.4 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 166 | 332
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Lumbar Spine Bone Mineral Density Percent Change From Baseline at Month 24
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 24 Months
Population: Randomized subjects who have a non-missing baseline and at least 1 non-missing postbaseline evaluation at or prior to month 24. LOCF was used as imputation method.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Denosumab 60 mg Q6M | Placebo
Number analyzed (Participants) | 163 | 163
Percent Change from Baseline | 6.5 [5.8 to 7.2] | -.6 [-1.2 to .1]
Statistical Analysis 1: Comparison: Denosumab 60 mg Q6M vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 7, 95% CI [6.2 to 7.8]

2. Secondary Outcome: Total Hip Bone Mineral Density Percent Change From Baseline at Month 24
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 24 Months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Denosumab 60 mg Q6M | Placebo
Number analyzed (Participants) | 163 | 163
Percent Change from Baseline | 3.4 [3.0 to 3.7] | -1.1 [-1.5 to -.8]

3. Secondary Outcome: Femoral Neck Bone Mineral Density Percent Change From Baseline at Month 24
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 24 Months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Denosumab 60 mg Q6M | Placebo
Number analyzed (Participants) | 163 | 163
Percent Change from Baseline | 2.8 [2.3 to 3.3] | -.9 [-1.4 to -.3]

4. Secondary Outcome: Trochanter Bone Mineral Density Percent Change From Baseline at Month 24
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 24 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Denosumab 60 mg Q6M | Placebo
Number analyzed (Participants) | 163 | 163
Percent Change from Baseline | 5.2 [4.7 to 5.6] | -.8 [-1.3 to -.3]

5. Secondary Outcome: Distal 1/3 Radius Bone Mineral Density Percent Change From Baseline at Month 24
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 24 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Denosumab 60 mg Q6M | Placebo
Number analyzed (Participants) | 156 | 156
Percent Change from Baseline | 1.4 [.9 to 1.9] | -2.1 [-2.6 to -1.6]

6. Secondary Outcome: Total Body (Without Head) Bone Mineral Density Percent Change From Baseline at Month 24
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry.
Time Frame: 24 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Denosumab 60 mg Q6M | Placebo
Number analyzed (Participants) | 156 | 154
Percent Change from Baseline | 2.4 [1.9 to 2.9] | -1.4 [-1.9 to -.8]

7. Secondary Outcome: Distal Radius Trabecular Volumetric Bone Mineral Density Percent Change From Baseline at Month 24
Description: Volumetric Bone Mineral Density Assessed by Quantitative Computerized Tomography (QCT).
Time Frame: 24 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Denosumab 60 mg Q6M | Placebo
Number analyzed (Participants) | 144 | 131
Percent Change from Baseline | 8.7 [3 to 14.4] | -.7 [-6.6 to 5.3]

8. Secondary Outcome: Distal Radius Cortical Volumetric Bone Mineral Density Percent Change From Baseline at Month 24
Description: Volumetric Bone Mineral Density Assessed by Quantitative Computerized Tomography (QCT).
Time Frame: 24 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Denosumab 60 mg Q6M | Placebo
Number analyzed (Participants) | 156 | 152
Percent Change from Baseline | .3 [-.1 to .8] | -1.4 [-1.8 to -.9]

9. Secondary Outcome: Distal Radius Total Volumetric Bone Mineral Density Percent Change From Baseline at Month 24
Description: Volumetric Bone Mineral Density Assessed by Quantitative Computerized Tomography (QCT).
Time Frame: 24 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change from Baseline
Arm/Group | Denosumab 60 mg Q6M | Placebo
Number analyzed (Participants) | 156 | 153
Percent Change from Baseline | .8 [0 to 1.6] | -1.9 [-2.6 to -1.1]

ADVERSE EVENTS:
Arm/Group | Placebo | Denosumab 60 mg Q6M
Serious Adverse Events (participants affected / at risk) | 9/165 | 18/164
Other Adverse Events (participants affected / at risk) | 157/165 | 156/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=165) | Denosumab 60 mg Q6M (N=164)
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 2
Lobar pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 3
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Facial palsy (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 1
Uterine perforation (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=165) | Denosumab 60 mg Q6M (N=164)
Abdominal pain (Gastrointestinal disorders) | 7 | 9
Constipation (Gastrointestinal disorders) | 8 | 18
Diarrhoea (Gastrointestinal disorders) | 7 | 14
Dyspepsia (Gastrointestinal disorders) | 10 | 9
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 9
Nausea (Gastrointestinal disorders) | 12 | 16
Fatigue (General disorders) | 12 | 7
Influenza (Infections and infestations) | 18 | 15
Nasopharyngitis (Infections and infestations) | 31 | 36
Sinusitis (Infections and infestations) | 17 | 10
Upper respiratory tract infection (Infections and infestations) | 22 | 19
Urinary tract infection (Infections and infestations) | 17 | 18
Procedural pain (Injury, poisoning and procedural complications) | 5 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 42 | 41
Back pain (Musculoskeletal and connective tissue disorders) | 33 | 33
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 24
Shoulder pain (Musculoskeletal and connective tissue disorders) | 10 | 17
Dizziness (Nervous system disorders) | 9 | 7
Headache (Nervous system disorders) | 19 | 26
Hypoaesthesia (Nervous system disorders) | 9 | 5
Depression (Psychiatric disorders) | 6 | 10
Insomnia (Psychiatric disorders) | 15 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 11
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 15
Rash (Skin and subcutaneous tissue disorders) | 5 | 14
Hypertension (Vascular disorders) | 14 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.